CLINICAL TRIAL: NCT00899587
Title: Evaluation of the Effects of Oxygen Therapy and Enalapril for Diabetic Macular Ischemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8753
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Diabetic Macular Ischemia
MeSH Terms: interventions — Enalapril; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxygen (Experimental)
  Interventions: Other: oxygen
- Enalapril (Experimental)
  Interventions: Drug: enalapril
- Control (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: enalapril — enalapril 5 mg every night
  Arms: Enalapril
Other: oxygen — oxygen 10 lit/min 1 hour twice a day at the first month, once a day at the second month and every other day at the third month
  Arms: Oxygen
Drug: placebo
  Arms: Control

SUMMARY:
In this study, patients were divided into 3 group with 35 cases including: 1.oxygen 2.enalapril 3.control.

In the beginning of the study, best corrected visual acuity (BCVA), uncorrected visual acuity (UCVA), and optical coherence tomography (OCT) were measured. Patients in the oxygen group were given oxygen 10 lit/min 1 hour twice a day at the first month, once a day at the second month and every other day at the third month. In the enalapril group, patients were given enalapril 5 mg every night and placebo was given for the patients in third group. At the end of first month the patients' vision was checked again and at the the end of the third month the first physical examinations were performed. In the first group, arterial blood gas (ABG) was taken before and after oxygen therapy as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetic macular ischemia

Exclusion Criteria:

* HTN > 1140/90 or HTN controlled by ACE inhibitors
* FBS > 200
* Severe anemia, COPD, cataract, HRPDR and diffuse macular edema

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran